CLINICAL TRIAL: NCT04646954
Title: DNA Methylation Testing for the Screening of Uterine Cervical Lesion: A Multicenter, Prospective Cohort Study
Brief Title: DNA Methylation Testing for the Screening of Uterine Cervical Lesion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METHY3
Record Dates: First submitted 2020-11-25; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia; DNA Methylation; High-risk Human Papillomavirus; Cytology
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: All eligible participants accept DNA methylation testing, with cytology and/or hrHPV assay in a hospital-based community。
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All eligible participants are included in the study group
  Interventions: Diagnostic Test: Host DNA methylation testing; Diagnostic Test: Cervical cytology and/or high-risk human papillomavirus assays

INTERVENTIONS:
Diagnostic Test: Host DNA methylation testing — Host EPB41L3, JAM3 and PAX1 methylation testing by cytology sample
Diagnostic Test: Cervical cytology and/or high-risk human papillomavirus assays — Cervical cytology and/or high-risk human papillomavirus assays

SUMMARY:
In our published work, host DNA methylation testing has been proved to be sensitive and specific to cervical intraepithelial neoplasia (CIN) 2 or more severe lesions (CIN2+). Its screening effects are independent of high-risk human papillomavirus (hrHPV) status. Based on the results of training and validation sets of our previous work, we perform this multicenter, prospective cohort study in unselected participants asking for cervical cancer screening in a hospital-based community. All eligible participants accept DNA methylation testing, with cytology and/or hrHPV assay. The primary endpoint is the diagnostic accuracy of DNA methylation compared with cytology and/or hrHPV status based on histology results. The accuracy analysis includes sensitivity, specificity, negative predictive value and positive predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years or older
* Signed an approved informed consents
* Feasible to be followed up
* Available residual cytology samples for methylation analysis

Exclusion Criteria:

* Without history of cervical disease, including cervical intraepithelial neoplasia (CIN) 2 or more severe lesions (CIN2+)
* No requirement of cervical cancer screening of cytology or high-risk human papillomavirus

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2022-11-26 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Two years
  The accuracy analysis includes sensitivity, specificity, negative predictive value and positive predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China